CLINICAL TRIAL: NCT02043496
Title: Integrative Cognitive-Affective Therapy for Binge Eating Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Neuropsychiatric Research Institute, Fargo, North Dakota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: PSYCH-2016-22310
Record Dates: First submitted 2014-01-14; First posted 2014-01-23 (Estimated); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Binge Eating Disorder
Keywords: Binge Eating Disorder; Binge Eating; Eating Disorders; Obesity; Psychotherapy; Cognitive Behavioral Therapy
MeSH Terms: conditions — Binge-Eating Disorder; Bulimia; Feeding and Eating Disorders; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CBT-Guided Self Help (Experimental): Integrative Cognitive-Affective Therapy CBT-Guided Self Help
  Interventions: Behavioral: CBT-Guided Self Help
- Integrative Cognitive-Affective Therapy (Experimental): Integrative Cognitive-Affective Therapy is a psychotherapy treatment for binge eating that focuses on changing behaviors, feelings, thoughts, and relationships
  Interventions: Behavioral: Integrative Cognitive-Affective Therapy

INTERVENTIONS:
Behavioral: Integrative Cognitive-Affective Therapy — Integrative Cognitive-Affective Therapy is a psychotherapy treatment for binge eating that focuses on changing behaviors, feelings, thoughts, and relationships
  Arms: Integrative Cognitive-Affective Therapy
Behavioral: CBT-Guided Self Help — CBT-Guided Self Help focuses on changing behavior patterns through the use of reading and homework assignments along with sessions with a therapist.
  Arms: CBT-Guided Self Help

SUMMARY:
The purpose of the study is to test a newly developed individual psychotherapy treatment for binge eating disorder in adults. This treatment is a type of individual psychotherapy called Integrative Cognitive-Affective Therapy (ICAT) that focuses on helping people change their behaviors, feelings, thoughts about themselves, and relationships. This new treatment is being compared to an existing treatment called Cognitive-Behavior Therapy-Guided Self Help (CBTgsh), which focuses on changing behavior patterns through the use of reading and homework assignments along with sessions with a therapist. The primary hypothesis of this investigation is that ICAT will be associated with greater reductions in binge eating at end of treatment and follow-up compared to CBTgsh.

ELIGIBILITY:
Inclusion Criteria:

* Binge eating disorder (DSM-5)

Exclusion Criteria:

* History of gastric bypass surgery
* Medical condition acutely affecting eating and/or weight
* Current medical and/or psychiatric instability (e.g., acute suicidality)
* Psychosis and/or bipolar disorder
* Severe cognitive impairment or developmental disability
* Inability to read English
* Current substance use disorder
* Current participation in psychotherapy and/or commercial weight loss program
* Change in dosage and/or frequency of psychotropic medication in the past 6 weeks
* Pregnant or breast feeding
* BMI < 21

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Binge Eating Episode Frequency (Eating Disorder Examination) | 17 Weeks and 6-month Follow-up
  Frequency of binge eating as measured by the Eating Disorder Examination

SECONDARY OUTCOMES:
Global Eating Disorder Symptoms (EDE) | 17 Weeks and 6-month follow-up
  Global Eating Disorder Symptoms as measured by the Eating Disorder Examination
Symptoms of Depression (BDI) | 17 Weeks and 6-month follow-up
  Symptoms of Depression as measured by the Beck Depression Inventory
Symptoms of Anxiety (STAI) | 17 Weeks and 6-month Follow-up
  Symptoms of Anxiety as measured by the State-Trait Anxiety Inventory
Self-Esteem (RSEQ) | 17 Weeks and 6-month Follow-up
  Self-esteem as measured by the Rosenberg Self-Esteem Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Carol B Peterson, PhD, Principal Investigator — University of Minnesota; Stephen A Wonderlich, PhD, Principal Investigator — Neuropsychiatric Research Institute/University of North Dakota
Locations (2):
- United States (2):
  - University of Minnesota, Minneapolis, Minnesota
  - Neuropsychiatric Research Institute, Fargo, North Dakota

REFERENCES:
- [Derived] Peterson CB, Engel SG, Crosby RD, Strauman T, Smith TL, Klein M, Crow SJ, Mitchell JE, Erickson A, Cao L, Bjorlie K, Wonderlich SA. Comparing integrative cognitive-affective therapy and guided self-help cognitive-behavioral therapy to treat binge-eating disorder using standard and naturalistic momentary outcome measures: A randomized controlled trial. Int J Eat Disord. 2020 Sep;53(9):1418-1427. doi: 10.1002/eat.23324. Epub 2020 Jun 25. PMID 32583478